CLINICAL TRIAL: NCT02990793
Title: A Prospective, Double Blind, Randomized, Sham-Controlled, Clinical Trial to Evaluate The Safety And Efficacy Of Biometrics-Guided Magnetic EEG Resonance Therapy (MeRT) Treatment Of Post-Traumatic Stress Disorder
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of MeRT Treatment in Post-Traumatic Stress Disorder
Acronym: MeRT-005-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Collaborators: Texas A&M University (Other); GilpinPhillips BIOMED, LLC (Unknown); Peachtree BioResearch Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MeRT-005-B
Record Dates: First submitted 2016-11-10; First posted 2016-12-13 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: PostTraumatic Stress Disorder; Traumatic Brain Injury; Postconcussive Symptoms
Keywords: PTSD; Concussion; TBI; TMS; Post Traumatic Stress Disorder; Posttraumatic Stress Disorder; Post-traumatic Stress Disorder; MERT; rTMS; Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active MeRT Treatment (Active Comparator): Active treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 5 weeks.
  Interventions: Device: Active MeRT Treatment
- Sham MeRT Treatment (Sham Comparator): Sham treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 5 weeks.
  Interventions: Device: Sham MeRT Treatment

INTERVENTIONS:
Device: Active MeRT Treatment — A personalized biometrics-guided protocol known as magnetic EEG/ECG resonance therapy (MeRT) treatment that is tailored specifically to each participant's EEG intrinsic alpha frequency (IAF). rTMS is applied at the participant's IAF.
  Other Names: rTMS Active Stimulator
  Arms: Active MeRT Treatment
Device: Sham MeRT Treatment — rTMS coil does not emit magnetic stimulation.
  Other Names: rTMS Sham Stimulator
  Arms: Sham MeRT Treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of individualized, Biometrics-guided Magnetic e-Resonance Therapy (MeRT) treatment of Post-Traumatic Stress Disorder

DETAILED DESCRIPTION:
MERT-005-B is a prospective, double blind, randomized, sham-controlled, parallel group, stratified, adaptive clinical trial designed to evaluate the efficacy of EEG-guided MeRT in persons with Post-Traumatic Stress Disorder

A total of 152 participants will be randomized in the Test Phase, and a group-sequential approach to efficacy monitoring by the Data and Safety Monitoring Board (DSMB).

A Pilot Phase was completed in which 74 participants were randomized. The Pilot Phase data will be used for confirming the safety of MeRT. For the Test Phase, eligible participants will be randomly assigned to either MeRT or Sham MeRT treatment groups in a 1:1 allocation ratio, with stratification on recruitment site and two levels of PPCS co-morbidity (+/-).

Initial eligibility evaluation and data collection will occur at the Screening Visit (SC). Following the SC visit, there will be a 5-week treatment period in which active or sham investigative treatment will be administered during daily weekday visits to the study site. Participants who received sham treatment and who continue to be eligible will be offered up to 25 active MeRT study treatments as part of Open Label Enrollment.

Main study outcomes will be collected at the second follow-up visit (F2) at the conclusion of the 5-week treatment period. An abbreviated data collection visit will occur during the third treatment week (the F1 follow-up visit). Additional follow up visits will occur 90 days after the first day of study treatment.

Participants, clinicians, and all personnel who participate in evaluation will be blind to study treatment group assignment.

The first phase of this trial was conducted in partnership with the United States Special Operations Command (USSOCOM) and the Henry Jackson Foundation.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all inclusion criteria to qualify for enrollment in the study:

1. Willing and able to consent to participate in the study
2. Age 18 - 65 years
3. Diagnosis of PTSD according to DSM-V criteria via CAPS-5
4. Onset of symptoms meeting the DSM-5 criteria for PTSD symptoms persisting for a minimum of 6 months prior to the Screening Visit
5. Minimum PCL-5 score of 30

Exclusion Criteria

Participants will be excluded from study participation if one or more of the following exclusion criteria apply:

1. Index trauma occurred before the age of 16 years
2. History of open skull injury
3. History of a neurological disorder including, but not limited to:

   * Seizure disorder
   * Any condition likely to be associated with increased intracranial pressure
   * Space occupying brain lesion
4. History of cerebrovascular accident
5. History of cerebral aneurysm
6. EEG abnormalities that indicate risk of seizure, i.e., abnormal focal or general slowing, or ictal spikes, during the EEG recording
7. Inability to calculate the EEG intrinsic alpha frequency at Screening
8. Participation in any interventional research protocol within 3 months prior to the Screening Visit
9. History of any type of ECT, rTMS, or MeRT treatment
10. Treated within 30 days of the Screening Visit with any antipsychotic medication
11. Treated within 30 days of the Screening Visit with any benzodiazepine or anticonvulsant medications
12. Current treatment with any restricted concomitant medication (i.e., NDRI, SSRI, SNRI, or QBDZ) that has not been stable for the preceding 60 days at the time of the Screening Visit
13. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within the head, excluding the mouth, or on the head, that cannot be safely removed
14. Biomedical devices, including those not in or on the head, that are either implanted or not safe to remove, that may be affected by the magnetic field of the stimulator (e.g., cardiac pacemaker, cardioverter defibrillator (ICD), or medication dispensing device)
15. Clinically significant medical illness or condition, including, but not limited to, any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunction, or chronic excessive alcohol consumption, that in the Investigator's judgment might pose a potential safety risk to the participant or limit the interpretation of trial results
16. Pregnant, or female unwilling to use effective birth control during the course of the trial
17. Plan to move away from the area, or knowledge that there will be an absence from the area, within 80 days following the Screening Visit (inclusive)
18. Unwilling or unable to adhere to the study treatment, data collection schedule, or study procedures, or any condition, including inability to communicate in English, which in the judgment of the Investigator might prevent the participant from completing the study, render study results uninterpretable, or represent an unacceptable safety risk to the participant or study personnel that is not otherwise listed in exclusion criteria.
19. Clinically significant psychopathology, including, but not limited to, schizophrenia or bipolar disorder, or other psychiatric disorder that in the Investigator's judgment might pose a potential safety risk to the participant, or limit the interpretation of trial results
20. An elevated risk of suicide or violence to others
21. Current psychotherapeutic treatment, expected to continue throughout the trial, that was begun in the preceding 60 days at the time of the Screening Visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptoms | Five weeks
  Change in PTSD symptoms as measured by the PTSD Checklist-5 (PCL-5).

OTHER OUTCOMES:
Safety Outcomes - Incidents and types of adverse events | Approximately 3 months
  Number and type of Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ramos, MD,PhD, Principal Investigator — Texas A&M University; Adele Gilpin, PhD,JD, Study Chair — GilpinPhillips BIOMED, LLC
Locations (8):
- United States (8):
  - BrainHealth Solutions, Costa Mesa, California
  - VA Long Beach Healthcare System, Long Beach, California
  - SoCal Neuroscience Research Unit, San Diego, California
  - UNC Rex Hospital, Raleigh, North Carolina
  - Columbus Brain Research Center, Columbus, Ohio
  - Center for Interventional Pain and Spine, Bryn Mawr, Pennsylvania
  - Texas A&M Research Center, Plano, Texas
  - Seattle Neuropsychiatric Treatment Center (Seattle NTC), Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abelson JL, Curtis GC, Sagher O, Albucher RC, Harrigan M, Taylor SF, Martis B, Giordani B. Deep brain stimulation for refractory obsessive-compulsive disorder. Biol Psychiatry. 2005 Mar 1;57(5):510-6. doi: 10.1016/j.biopsych.2004.11.042. PMID 15737666
- [Background] Achard S, Delon-Martin C, Vertes PE, Renard F, Schenck M, Schneider F, Heinrich C, Kremer S, Bullmore ET. Hubs of brain functional networks are radically reorganized in comatose patients. Proc Natl Acad Sci U S A. 2012 Dec 11;109(50):20608-13. doi: 10.1073/pnas.1208933109. Epub 2012 Nov 26. PMID 23185007
- [Background] ACRM: Mild Traumatic Brain Injury Committee. (1993). Definition of mild traumatic brain injury. J Head Trauma Rehabil, 8, 86-87.
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders (5th ed.). Washington, DC: American Psychiatric Publishing.
- [Background] American Psychiatric Association. (2013). PTSD: National Center for PTSD. Retrieved October 12, 2020, from U.S. Department of Veterans Affairs: https://www.ptsd.va.gov/professional/treat/essentials/
- [Background] American Psychiatric Association Task Force on DSM-IV. (2000). Diagnostic and statistical manual of mental disorders: DSM-IV-TR. 4th ed. Washington, DC: American Psychiatric Association.
- [Background] Anderson B, Mishory A, Nahas Z, Borckardt JJ, Yamanaka K, Rastogi K, George MS. Tolerability and safety of high daily doses of repetitive transcranial magnetic stimulation in healthy young men. J ECT. 2006 Mar;22(1):49-53. doi: 10.1097/00124509-200603000-00011. PMID 16633208
- [Background] Arciniegas DB, Silver JM. Regarding the search for a unified definition of mild traumatic brain injury. Brain Inj. 2001 Jul;15(7):649-52. doi: 10.1080/02699050010019800. No abstract available. PMID 11429094
- [Background] Bae EH, Schrader LM, Machii K, Alonso-Alonso M, Riviello JJ Jr, Pascual-Leone A, Rotenberg A. Safety and tolerability of repetitive transcranial magnetic stimulation in patients with epilepsy: a review of the literature. Epilepsy Behav. 2007 Jun;10(4):521-8. doi: 10.1016/j.yebeh.2007.03.004. Epub 2007 May 9. PMID 17493877
- [Background] Bang, H., Flaherty, S. P., Kolahi, J., & Park, J. (2010). Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol. Clinical Research and Regulatory Affairs, 27(2), 42 - 51.
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Benjet C, Bromet E, Karam EG, Kessler RC, McLaughlin KA, Ruscio AM, Shahly V, Stein DJ, Petukhova M, Hill E, Alonso J, Atwoli L, Bunting B, Bruffaerts R, Caldas-de-Almeida JM, de Girolamo G, Florescu S, Gureje O, Huang Y, Lepine JP, Kawakami N, Kovess-Masfety V, Medina-Mora ME, Navarro-Mateu F, Piazza M, Posada-Villa J, Scott KM, Shalev A, Slade T, ten Have M, Torres Y, Viana MC, Zarkov Z, Koenen KC. The epidemiology of traumatic event exposure worldwide: results from the World Mental Health Survey Consortium. Psychol Med. 2016 Jan;46(2):327-43. doi: 10.1017/S0033291715001981. Epub 2015 Oct 29. PMID 26511595
- [Background] Bikson M, Hanlon CA, Woods AJ, Gillick BT, Charvet L, Lamm C, Madeo G, Holczer A, Almeida J, Antal A, Ay MR, Baeken C, Blumberger DM, Campanella S, Camprodon JA, Christiansen L, Loo C, Crinion JT, Fitzgerald P, Gallimberti L, Ghobadi-Azbari P, Ghodratitoostani I, Grabner RH, Hartwigsen G, Hirata A, Kirton A, Knotkova H, Krupitsky E, Marangolo P, Nakamura-Palacios EM, Potok W, Praharaj SK, Ruff CC, Schlaug G, Siebner HR, Stagg CJ, Thielscher A, Wenderoth N, Yuan TF, Zhang X, Ekhtiari H. Guidelines for TMS/tES clinical services and research through the COVID-19 pandemic. Brain Stimul. 2020 Jul-Aug;13(4):1124-1149. doi: 10.1016/j.brs.2020.05.010. Epub 2020 May 12. PMID 32413554
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Bjork JM, Burroughs TK, Franke LM, Pickett TC, Johns SE, Moeller FG, Walker WC. Laboratory impulsivity and depression in blast-exposed military personnel with post-concussion syndrome. Psychiatry Res. 2016 Dec 30;246:321-325. doi: 10.1016/j.psychres.2016.10.008. Epub 2016 Oct 7. PMID 27750113
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Blyth BJ, Bazarian JJ. Traumatic alterations in consciousness: traumatic brain injury. Emerg Med Clin North Am. 2010 Aug;28(3):571-94. doi: 10.1016/j.emc.2010.03.003. PMID 20709244
- [Background] Bogner J, Corrigan JD. Reliability and predictive validity of the Ohio State University TBI identification method with prisoners. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):279-91. doi: 10.1097/HTR.0b013e3181a66356. PMID 19625867
- [Background] Bonita JD, Ambolode LC 2nd, Rosenberg BM, Cellucci CJ, Watanabe TA, Rapp PE, Albano AM. Time domain measures of inter-channel EEG correlations: a comparison of linear, nonparametric and nonlinear measures. Cogn Neurodyn. 2014 Feb;8(1):1-15. doi: 10.1007/s11571-013-9267-8. Epub 2013 Sep 4. PMID 24465281
- [Background] Boutros NN, Gueorguieva R, Hoffman RE, Oren DA, Feingold A, Berman RM. Lack of a therapeutic effect of a 2-week sub-threshold transcranial magnetic stimulation course for treatment-resistant depression. Psychiatry Res. 2002 Dec 30;113(3):245-54. doi: 10.1016/s0165-1781(02)00267-6. PMID 12559481
- [Background] Bradley KA, Bush KR, Epler AJ, Dobie DJ, Davis TM, Sporleder JL, Maynard C, Burman ML, Kivlahan DR. Two brief alcohol-screening tests From the Alcohol Use Disorders Identification Test (AUDIT): validation in a female Veterans Affairs patient population. Arch Intern Med. 2003 Apr 14;163(7):821-9. doi: 10.1001/archinte.163.7.821. PMID 12695273
- [Background] Breslau N, Davis GC, Andreski P, Peterson E. Traumatic events and posttraumatic stress disorder in an urban population of young adults. Arch Gen Psychiatry. 1991 Mar;48(3):216-22. doi: 10.1001/archpsyc.1991.01810270028003. PMID 1996917
- [Background] Breslau N. Outcomes of posttraumatic stress disorder. J Clin Psychiatry. 2001;62 Suppl 17:55-9. PMID 11495098
- [Background] Breslau N. The epidemiology of posttraumatic stress disorder: what is the extent of the problem? J Clin Psychiatry. 2001;62 Suppl 17:16-22. PMID 11495091
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carroll LJ, Cassidy JD, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Methodological issues and research recommendations for mild traumatic brain injury: the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):113-25. doi: 10.1080/16501960410023877. PMID 15083875
- [Background] Castellanos NP, Bajo R, Cuesta P, Villacorta-Atienza JA, Paul N, Garcia-Prieto J, Del-Pozo F, Maestu F. Alteration and reorganization of functional networks: a new perspective in brain injury study. Front Hum Neurosci. 2011 Sep 21;5:90. doi: 10.3389/fnhum.2011.00090. eCollection 2011. PMID 21960965
- [Background] Castellanos NP, Paul N, Ordonez VE, Demuynck O, Bajo R, Campo P, Bilbao A, Ortiz T, del-Pozo F, Maestu F. Reorganization of functional connectivity as a correlate of cognitive recovery in acquired brain injury. Brain. 2010 Aug;133(Pt 8):2365-81. doi: 10.1093/brain/awq174. PMID 20826433
- [Background] Caulfield KA. Is accelerated, high-dose theta burst stimulation a panacea for treatment-resistant depression? J Neurophysiol. 2020 Jan 1;123(1):1-3. doi: 10.1152/jn.00537.2019. Epub 2019 Sep 25. PMID 31553674
- [Background] Chen YH, DeMets DL, Lan KK. Increasing the sample size when the unblinded interim result is promising. Stat Med. 2004 Apr 15;23(7):1023-38. doi: 10.1002/sim.1688. PMID 15057876
- [Background] Comerchero MD, Polich J. P3a and P3b from typical auditory and visual stimuli. Clin Neurophysiol. 1999 Jan;110(1):24-30. doi: 10.1016/s0168-5597(98)00033-1. PMID 10348317
- [Background] CONSORT Group. (2010). CONSORT 2010. Retrieved January 13, 2016, from CONSORT Transparent Reporting of Trials: http://www.consort-statement.org/consort-2010
- [Background] Corlier J, Carpenter LL, Wilson AC, Tirrell E, Gobin AP, Kavanaugh B, Leuchter AF. The relationship between individual alpha peak frequency and clinical outcome with repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder (MDD). Brain Stimul. 2019 Nov-Dec;12(6):1572-1578. doi: 10.1016/j.brs.2019.07.018. Epub 2019 Jul 25. PMID 31378603
- [Background] Corrigan JD, Bogner J. Initial reliability and validity of the Ohio State University TBI Identification Method. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):318-29. doi: 10.1097/01.HTR.0000300227.67748.77. PMID 18025964
- [Background] Davidson JR, Hughes D, Blazer DG, George LK. Post-traumatic stress disorder in the community: an epidemiological study. Psychol Med. 1991 Aug;21(3):713-21. doi: 10.1017/s0033291700022352. PMID 1946860
- [Background] De Beaumont L, Mongeon D, Tremblay S, Messier J, Prince F, Leclerc S, Lassonde M, Theoret H. Persistent motor system abnormalities in formerly concussed athletes. J Athl Train. 2011 May-Jun;46(3):234-40. doi: 10.4085/1062-6050-46.3.234. PMID 21669091
- [Background] Department of Defense. (2011, November). Department of Defense Instruction 3216.02.
- [Background] Dhamne SC, Kothare RS, Yu C, Hsieh TH, Anastasio EM, Oberman L, Pascual-Leone A, Rotenberg A. A measure of acoustic noise generated from transcranial magnetic stimulation coils. Brain Stimul. 2014 May-Jun;7(3):432-4. doi: 10.1016/j.brs.2014.01.056. Epub 2014 Jan 29. PMID 24582370
- [Background] Di Stefano G, Bachevalier J, Levin HS, Song JX, Scheibel RS, Fletcher JM. Volume of focal brain lesions and hippocampal formation in relation to memory function after closed head injury in children. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):210-6. doi: 10.1136/jnnp.69.2.210. PMID 10896695
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Dupont, W. D., & Plummer, W. D. (1997). Power and Sample Size software. Controlled Clinical Trials, 18, 274.
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations for studies involving linear regression. Control Clin Trials. 1998 Dec;19(6):589-601. doi: 10.1016/s0197-2456(98)00037-3. PMID 9875838
- [Background] Eckberg, D. L. (2004). Correlations among heart rate variability components and autonomic mechanisms. In M. Malik, & J. A. Camm (Eds.), Dynamic Electrocardiology (pp. 31-39). Elmsford, NY, US: Blackwell/Futura.
- [Background] Evidence-based Synthesis Program (ESP) Center, Portland VA Medical Center. (2015, November). Systematic Review of Suicide Prevention in Veterans. Retrieved October 24, 2020, from U.S. Department of Veterans Affairs: https://www.hsrd.research.va.gov/publications/esp/SuicidePrevention-REPORT.pdf
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Garcia-Gonzalez MA, Fernandez-Chimeno M, Ferrer J, Escorihuela RM, Parrado E, Capdevila L, Benitez A, Angulo R, Rodriguez FA, Iglesias X, Bescos R, Marina M, Padulles JM, Ramos-Castro J. New indices for quantification of the power spectrum of heart rate variability time series without the need of any frequency band definition. Physiol Meas. 2011 Aug;32(8):995-1009. doi: 10.1088/0967-3334/32/8/001. Epub 2011 Jun 7. PMID 21654027
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434
- [Background] George MS, Wassermann EM, Williams WA, Steppel J, Pascual-Leone A, Basser P, Hallett M, Post RM. Changes in mood and hormone levels after rapid-rate transcranial magnetic stimulation (rTMS) of the prefrontal cortex. J Neuropsychiatry Clin Neurosci. 1996 Spring;8(2):172-80. doi: 10.1176/jnp.8.2.172. PMID 9081553
- [Background] Gersons BP, Carlier IV. Post-traumatic stress disorder: the history of a recent concept. Br J Psychiatry. 1992 Dec;161:742-8. doi: 10.1192/bjp.161.6.742. PMID 1483159
- [Background] Geuze E, Vermetten E, Bremner JD. MR-based in vivo hippocampal volumetrics: 2. Findings in neuropsychiatric disorders. Mol Psychiatry. 2005 Feb;10(2):160-84. doi: 10.1038/sj.mp.4001579. PMID 15356639
- [Background] Gevins A, Cutillo B. Spatiotemporal dynamics of component processes in human working memory. Electroencephalogr Clin Neurophysiol. 1993 Sep;87(3):128-43. doi: 10.1016/0013-4694(93)90119-g. PMID 7691540
- [Background] Gondusky JS, Reiter MP. Protecting military convoys in Iraq: an examination of battle injuries sustained by a mechanized battalion during Operation Iraqi Freedom II. Mil Med. 2005 Jun;170(6):546-9. doi: 10.7205/milmed.170.6.546. PMID 16001610
- [Background] Gordon WA, Haddad L, Brown M, Hibbard MR, Sliwinski M. The sensitivity and specificity of self-reported symptoms in individuals with traumatic brain injury. Brain Inj. 2000 Jan;14(1):21-33. PMID 10670659
- [Background] Hardmeier M, Hatz F, Bousleiman H, Schindler C, Stam CJ, Fuhr P. Reproducibility of functional connectivity and graph measures based on the phase lag index (PLI) and weighted phase lag index (wPLI) derived from high resolution EEG. PLoS One. 2014 Oct 6;9(10):e108648. doi: 10.1371/journal.pone.0108648. eCollection 2014. PMID 25286380
- [Background] Helzer JE, Robins LN, McEvoy L. Post-traumatic stress disorder in the general population. Findings of the epidemiologic catchment area survey. N Engl J Med. 1987 Dec 24;317(26):1630-4. doi: 10.1056/NEJM198712243172604. PMID 3683502
- [Background] Herwig U, Fallgatter AJ, Hoppner J, Eschweiler GW, Kron M, Hajak G, Padberg F, Naderi-Heiden A, Abler B, Eichhammer P, Grossheinrich N, Hay B, Kammer T, Langguth B, Laske C, Plewnia C, Richter MM, Schulz M, Unterecker S, Zinke A, Spitzer M, Schonfeldt-Lecuona C. Antidepressant effects of augmentative transcranial magnetic stimulation: randomised multicentre trial. Br J Psychiatry. 2007 Nov;191:441-8. doi: 10.1192/bjp.bp.106.034371. PMID 17978325
- [Background] Hien DA, Jiang H, Campbell AN, Hu MC, Miele GM, Cohen LR, Brigham GS, Capstick C, Kulaga A, Robinson J, Suarez-Morales L, Nunes EV. Do treatment improvements in PTSD severity affect substance use outcomes? A secondary analysis from a randomized clinical trial in NIDA's Clinical Trials Network. Am J Psychiatry. 2010 Jan;167(1):95-101. doi: 10.1176/appi.ajp.2009.09091261. Epub 2009 Nov 16. PMID 19917596
- [Background] Hoge CW, Goldberg HM, Castro CA. Care of war veterans with mild traumatic brain injury--flawed perspectives. N Engl J Med. 2009 Apr 16;360(16):1588-91. doi: 10.1056/NEJMp0810606. No abstract available. PMID 19369664
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Hoge CW, Yehuda R, Castro CA, McFarlane AC, Vermetten E, Jetly R, Koenen KC, Greenberg N, Shalev AY, Rauch SA, Marmar CR, Rothbaum BO. Unintended Consequences of Changing the Definition of Posttraumatic Stress Disorder in DSM-5: Critique and Call for Action. JAMA Psychiatry. 2016 Jul 1;73(7):750-2. doi: 10.1001/jamapsychiatry.2016.0647. No abstract available. PMID 27224895
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Hunter AM, Minzenberg MJ, Cook IA, Krantz DE, Levitt JG, Rotstein NM, Chawla SA, Leuchter AF. Concomitant medication use and clinical outcome of repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder. Brain Behav. 2019 May;9(5):e01275. doi: 10.1002/brb3.1275. Epub 2019 Apr 2. PMID 30941915
- [Background] Ingebrigtsen T, Waterloo K, Marup-Jensen S, Attner E, Romner B. Quantification of post-concussion symptoms 3 months after minor head injury in 100 consecutive patients. J Neurol. 1998 Sep;245(9):609-12. doi: 10.1007/s004150050254. PMID 9758300
- [Background] International Committee Of Medical Journal Editors. [Recommendations for the conduct, reporting, editing and publication of scholarly work in medical journals (revised in January 2024): a Korean translation]. Ewha Med J. 2024 Oct;47(4):e48. doi: 10.12771/emj.2024.e48. Epub 2024 Oct 31. No abstract available. Korean. PMID 40704003
- [Background] James KE, Bloch DA, Lee KK, Kraemer HC, Fuller RK. An index for assessing blindness in a multi-centre clinical trial: disulfiram for alcohol cessation--a VA cooperative study. Stat Med. 1996 Jul 15;15(13):1421-34. doi: 10.1002/(SICI)1097-0258(19960715)15:133.0.CO;2-H. PMID 8841652
- [Background] Janicak PG, O'Reardon JP, Sampson SM, Husain MM, Lisanby SH, Rado JT, Heart KL, Demitrack MA. Transcranial magnetic stimulation in the treatment of major depressive disorder: a comprehensive summary of safety experience from acute exposure, extended exposure, and during reintroduction treatment. J Clin Psychiatry. 2008 Feb;69(2):222-32. doi: 10.4088/jcp.v69n0208. PMID 18232722
- [Background] Jin Y, Phillips B. A pilot study of the use of EEG-based synchronized Transcranial Magnetic Stimulation (sTMS) for treatment of Major Depression. BMC Psychiatry. 2014 Jan 18;14:13. doi: 10.1186/1471-244X-14-13. PMID 24438321
- [Background] Jin Y, Kemp AS, Huang Y, Thai TM, Liu Z, Xu W, He H, Potkin SG. Alpha EEG guided TMS in schizophrenia. Brain Stimul. 2012 Oct;5(4):560-8. doi: 10.1016/j.brs.2011.09.005. Epub 2011 Oct 6. PMID 22019083
- [Background] Jin Y, Potkin SG, Kemp AS, Huerta ST, Alva G, Thai TM, Carreon D, Bunney WE Jr. Therapeutic effects of individualized alpha frequency transcranial magnetic stimulation (alphaTMS) on the negative symptoms of schizophrenia. Schizophr Bull. 2006 Jul;32(3):556-61. doi: 10.1093/schbul/sbj020. Epub 2005 Oct 27. PMID 16254067
- [Background] Johns, M. (n.d.). About the ESS. Retrieved October 23, 2020, from The Epworth Sleepiness Scale: https://epworthsleepinessscale.com/about-the-ess/
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Keane, T. M., Fairbank, J. A., Caddel, J. M., Zimering, R. T., Taylor, K. L., & Mora, C. A. (1989). Clinical Evaluation of a Measure to Assess Combat Exposure. Psychological Assessment, 1(1), 53 - 55.
- [Background] Kehle SM, Reddy MK, Ferrier-Auerbach AG, Erbes CR, Arbisi PA, Polusny MA. Psychiatric diagnoses, comorbidity, and functioning in National Guard troops deployed to Iraq. J Psychiatr Res. 2011 Jan;45(1):126-32. doi: 10.1016/j.jpsychires.2010.05.013. Epub 2010 Jun 11. PMID 20541221
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Kessler RC. Posttraumatic stress disorder: the burden to the individual and to society. J Clin Psychiatry. 2000;61 Suppl 5:4-12; discussion 13-4. PMID 10761674
- [Background] Kilpatrick DG, Resnick HS, Milanak ME, Miller MW, Keyes KM, Friedman MJ. National estimates of exposure to traumatic events and PTSD prevalence using DSM-IV and DSM-5 criteria. J Trauma Stress. 2013 Oct;26(5):537-47. doi: 10.1002/jts.21848. PMID 24151000
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Klimesch W. An algorithm for the EEG frequency architecture of consciousness and brain body coupling. Front Hum Neurosci. 2013 Nov 12;7:766. doi: 10.3389/fnhum.2013.00766. eCollection 2013. No abstract available. PMID 24273507
- [Background] Kobayashi B, Cook IA, Hunter AM, Minzenberg MJ, Krantz DE, Leuchter AF. Can neurophysiologic measures serve as biomarkers for the efficacy of repetitive transcranial magnetic stimulation treatment of major depressive disorder? Int Rev Psychiatry. 2017 Apr;29(2):98-114. doi: 10.1080/09540261.2017.1297697. Epub 2017 Mar 31. PMID 28362541
- [Background] Kroenke, K., & Spitzer, R. L. (2002, September). The PHQ-9: A New Depression Diagnostic and Severity Measure. Psychiatric Annals, 32(9), 1 - 7.
- [Background] Lerner AJ, Wassermann EM, Tamir DI. Seizures from transcranial magnetic stimulation 2012-2016: Results of a survey of active laboratories and clinics. Clin Neurophysiol. 2019 Aug;130(8):1409-1416. doi: 10.1016/j.clinph.2019.03.016. Epub 2019 Apr 6. PMID 31104898
- [Background] Leuchter AF, Cook IA, Jin Y, Phillips B. The relationship between brain oscillatory activity and therapeutic effectiveness of transcranial magnetic stimulation in the treatment of major depressive disorder. Front Hum Neurosci. 2013 Feb 26;7:37. doi: 10.3389/fnhum.2013.00037. eCollection 2013. PMID 23550274
- [Background] Ling G, Bandak F, Armonda R, Grant G, Ecklund J. Explosive blast neurotrauma. J Neurotrauma. 2009 Jun;26(6):815-25. doi: 10.1089/neu.2007.0484. PMID 19397423
- [Background] Liu Y, Liang M, Zhou Y, He Y, Hao Y, Song M, Yu C, Liu H, Liu Z, Jiang T. Disrupted small-world networks in schizophrenia. Brain. 2008 Apr;131(Pt 4):945-61. doi: 10.1093/brain/awn018. Epub 2008 Feb 25. PMID 18299296
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Loo C, Sachdev P, Elsayed H, McDarmont B, Mitchell P, Wilkinson M, Parker G, Gandevia S. Effects of a 2- to 4-week course of repetitive transcranial magnetic stimulation (rTMS) on neuropsychologic functioning, electroencephalogram, and auditory threshold in depressed patients. Biol Psychiatry. 2001 Apr 1;49(7):615-23. doi: 10.1016/s0006-3223(00)00996-3. PMID 11297719
- [Background] Lopes da Silva, F. (2005(a)). EEG analysis: theory and practice. In E. Niedermeyer, & F. Lopes da Silva (Eds.), Electroencephalography; Basic Principles, Clinical Applications and Related Fields (pp. 1199-1231). Philadelphia, PA, USA: Lippincott, Williams and Wilkins.
- [Background] Lopes da Silva, F. (2005(b)). Events-related potentials: methodology and quantification. In E. Niedermeyer, & F. Lopes da Silva, Electroencephalography: Basic Principles, Clinical Applications and Related Fields (pp. 991-1001). Philadelphia, Pennsylvania, US: Lippincott, Williams and Wilkins.
- [Background] Luck, S. J. (2005). An Introduction to the Event-Related Potential Technique. Cambridge, MA, US: MIT Press.
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] Madulara, M. D., Francisco, P. A., Nawang, S., Arogancia, D. C., Cellucci, C. J., Rapp, P. E., & Albano, A. M. (2012). EEG transfer entropy tracks changes of information transfer on the onset of vision. International Journal of Modern Physics, 17, 9-18.
- [Background] Mayer G, Aviram S, Walter G, Levkovitz Y, Bloch Y. Long-term follow-up of adolescents with resistant depression treated with repetitive transcranial magnetic stimulation. J ECT. 2012 Jun;28(2):84-6. doi: 10.1097/YCT.0b013e318238f01a. PMID 22531199
- [Background] Mayo Clinic Staff. (n.d.). Post-concussion syndrome. Retrieved September 15, 2015, from Mayo Clinic: http://www.mayoclinic.org/diseases-conditions/post-concussion-syndrome/basics/treatment/con-20032705
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Background] McCrea, M, ed; American Academy of Clinical Neuropsychology. (2008). Mild traumatic brain injury and postconcussion syndrome: the new evidence base for diagnosis and treatment. Oxford; New York: Oxford University Press.
- [Background] McGough JJ, Sturm A, Cowen J, Tung K, Salgari GC, Leuchter AF, Cook IA, Sugar CA, Loo SK. Double-Blind, Sham-Controlled, Pilot Study of Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2019 Apr;58(4):403-411.e3. doi: 10.1016/j.jaac.2018.11.013. Epub 2019 Jan 28. PMID 30768393
- [Background] Menon DK, Schwab K, Wright DW, Maas AI; Demographics and Clinical Assessment Working Group of the International and Interagency Initiative toward Common Data Elements for Research on Traumatic Brain Injury and Psychological Health. Position statement: definition of traumatic brain injury. Arch Phys Med Rehabil. 2010 Nov;91(11):1637-40. doi: 10.1016/j.apmr.2010.05.017. PMID 21044706
- [Background] Miller, M. W., Wolf, E. J., Kilpatrick, D., Resnick, H., Marx, B. P., Holowka, D. W., . . . Friedman, M. J. (2012). The Prevalence and Latent Structure of Proposed DSM-5 Posttraumatic Stress Disorder Symptoms in U.S. National and Veteran Samples. Psychological Trauma: Theory, Research, Practice, and Policy. doi:10.1037/a0029730
- [Background] Mittenberg W, Strauman S. Diagnosis of mild head injury and the postconcussion syndrome. J Head Trauma Rehabil. 2000 Apr;15(2):783-91. doi: 10.1097/00001199-200004000-00003. PMID 10739967
- [Background] Mittenberg W, Wittner MS, Miller LJ. Postconcussion syndrome occurs in children. Neuropsychology. 1997 Jul;11(3):447-52. doi: 10.1037//0894-4105.11.3.447. PMID 9223149
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Nintendo of America Inc. (2015). Nintendo Gameboy Manual. Redmond, WA.
- [Background] Okie S. Traumatic brain injury in the war zone. N Engl J Med. 2005 May 19;352(20):2043-7. doi: 10.1056/NEJMp058102. No abstract available. PMID 15901856
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Owen AM, McMillan KM, Laird AR, Bullmore E. N-back working memory paradigm: a meta-analysis of normative functional neuroimaging studies. Hum Brain Mapp. 2005 May;25(1):46-59. doi: 10.1002/hbm.20131. PMID 15846822
- [Background] Pascual-Leone A, Catala MD, Pascual-Leone Pascual A. Lateralized effect of rapid-rate transcranial magnetic stimulation of the prefrontal cortex on mood. Neurology. 1996 Feb;46(2):499-502. doi: 10.1212/wnl.46.2.499. PMID 8614521
- [Background] Pascual-Leone A, Cohen LG, Shotland LI, Dang N, Pikus A, Wassermann EM, Brasil-Neto JP, Valls-Sole J, Hallett M. No evidence of hearing loss in humans due to transcranial magnetic stimulation. Neurology. 1992 Mar;42(3 Pt 1):647-51. doi: 10.1212/wnl.42.3.647. PMID 1549231
- [Background] Pascual-Leone A, Houser CM, Reese K, Shotland LI, Grafman J, Sato S, Valls-Sole J, Brasil-Neto JP, Wassermann EM, Cohen LG, et al. Safety of rapid-rate transcranial magnetic stimulation in normal volunteers. Electroencephalogr Clin Neurophysiol. 1993 Apr;89(2):120-30. doi: 10.1016/0168-5597(93)90094-6. PMID 7683602
- [Background] Perera T, George MS, Grammer G, Janicak PG, Pascual-Leone A, Wirecki TS. The Clinical TMS Society Consensus Review and Treatment Recommendations for TMS Therapy for Major Depressive Disorder. Brain Stimul. 2016 May-Jun;9(3):336-346. doi: 10.1016/j.brs.2016.03.010. Epub 2016 Mar 16. PMID 27090022
- [Background] Peskind ER, Petrie EC, Cross DJ, Pagulayan K, McCraw K, Hoff D, Hart K, Yu CE, Raskind MA, Cook DG, Minoshima S. Cerebrocerebellar hypometabolism associated with repetitive blast exposure mild traumatic brain injury in 12 Iraq war Veterans with persistent post-concussive symptoms. Neuroimage. 2011 Jan;54 Suppl 1(Suppl 1):S76-82. doi: 10.1016/j.neuroimage.2010.04.008. Epub 2010 Apr 10. PMID 20385245
- [Background] Philip NS, Carpenter SL, Ridout SJ, Sanchez G, Albright SE, Tyrka AR, Price LH, Carpenter LL. 5Hz Repetitive transcranial magnetic stimulation to left prefrontal cortex for major depression. J Affect Disord. 2015 Nov 1;186:13-7. doi: 10.1016/j.jad.2014.12.024. Epub 2015 Jul 17. PMID 26210705
- [Background] Pinna GD, Maestri R, Torunski A, Danilowicz-Szymanowicz L, Szwoch M, La Rovere MT, Raczak G. Heart rate variability measures: a fresh look at reliability. Clin Sci (Lond). 2007 Aug;113(3):131-40. doi: 10.1042/CS20070055. PMID 17381425
- [Background] Polich J, Criado JR. Neuropsychology and neuropharmacology of P3a and P3b. Int J Psychophysiol. 2006 May;60(2):172-85. doi: 10.1016/j.ijpsycho.2005.12.012. Epub 2006 Feb 28. PMID 16510201
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Porta A, Bari V, Marchi A, De Maria B, Cysarz D, Van Leeuwen P, Takahashi AC, Catai AM, Gnecchi-Ruscone T. Complexity analyses show two distinct types of nonlinear dynamics in short heart period variability recordings. Front Physiol. 2015 Mar 10;6:71. doi: 10.3389/fphys.2015.00071. eCollection 2015. PMID 25806002
- [Background] Abdul Razak F, Jensen HJ. Quantifying 'causality' in complex systems: understanding transfer entropy. PLoS One. 2014 Jun 23;9(6):e99462. doi: 10.1371/journal.pone.0099462. eCollection 2014. PMID 24955766
- [Background] Regier DA, Narrow WE, Clarke DE, Kraemer HC, Kuramoto SJ, Kuhl EA, Kupfer DJ. DSM-5 field trials in the United States and Canada, Part II: test-retest reliability of selected categorical diagnoses. Am J Psychiatry. 2013 Jan;170(1):59-70. doi: 10.1176/appi.ajp.2012.12070999. PMID 23111466
- [Background] Richman JS, Moorman JR. Physiological time-series analysis using approximate entropy and sample entropy. Am J Physiol Heart Circ Physiol. 2000 Jun;278(6):H2039-49. doi: 10.1152/ajpheart.2000.278.6.H2039. PMID 10843903
- [Background] Roelofs CL, Krepel N, Corlier J, Carpenter LL, Fitzgerald PB, Daskalakis ZJ, Tendolkar I, Wilson A, Downar J, Bailey NW, Blumberger DM, Vila-Rodriguez F, Leuchter AF, Arns M. Individual alpha frequency proximity associated with repetitive transcranial magnetic stimulation outcome: An independent replication study from the ICON-DB consortium. Clin Neurophysiol. 2021 Feb;132(2):643-649. doi: 10.1016/j.clinph.2020.10.017. Epub 2020 Nov 10. PMID 33243617
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Runge J, Heitzig J, Marwan N, Kurths J. Quantifying causal coupling strength: a lag-specific measure for multivariate time series related to transfer entropy. Phys Rev E Stat Nonlin Soft Matter Phys. 2012 Dec;86(6 Pt 1):061121. doi: 10.1103/PhysRevE.86.061121. Epub 2012 Dec 17. PMID 23367907
- [Background] Sakkas P, Mihalopoulou P, Mourtzouhou P, Psarros C, Masdrakis V, Politis A, Christodoulou GN. Induction of mania by rTMS: report of two cases. Eur Psychiatry. 2003 Jun;18(4):196-8. doi: 10.1016/s0924-9338(03)00048-8. PMID 12814856
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Sigurdardottir S, Andelic N, Roe C, Jerstad T, Schanke AK. Post-concussion symptoms after traumatic brain injury at 3 and 12 months post-injury: a prospective study. Brain Inj. 2009 Jun;23(6):489-97. doi: 10.1080/02699050902926309. PMID 19484622
- [Background] Silver JM, McAllister TW. Forensic issues in the neuropsychiatric evaluation of the patient with mild traumatic brain injury. J Neuropsychiatry Clin Neurosci. 1997 Winter;9(1):102-13. doi: 10.1176/jnp.9.1.102. No abstract available. PMID 9017537
- [Background] Spencer, K. M. (2005). Averaging, detection and classification of single-trial ERPs. In T. M. Handy (Ed.), Event Related Potentials. A Methods Handbook (pp. 209-227). Cambridge, MA, US: MIT Press.
- [Background] Spoont M, Arbisi P, Fu S, Greer N, Kehle-Forbes S, Meis L, Rutks I, Wilt TJ. Screening for Post-Traumatic Stress Disorder (PTSD) in Primary Care: A Systematic Review [Internet]. Washington (DC): Department of Veterans Affairs (US); 2013 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK126691/ PMID 23487872
- [Background] Stein DJ, McLaughlin KA, Koenen KC, Atwoli L, Friedman MJ, Hill ED, Maercker A, Petukhova M, Shahly V, van Ommeren M, Alonso J, Borges G, de Girolamo G, de Jonge P, Demyttenaere K, Florescu S, Karam EG, Kawakami N, Matschinger H, Okoliyski M, Posada-Villa J, Scott KM, Viana MC, Kessler RC. DSM-5 and ICD-11 definitions of posttraumatic stress disorder: investigating "narrow" and "broad" approaches. Depress Anxiety. 2014 Jun;31(6):494-505. doi: 10.1002/da.22279. PMID 24894802
- [Background] Stein MB, McAllister TW. Exploring the convergence of posttraumatic stress disorder and mild traumatic brain injury. Am J Psychiatry. 2009 Jul;166(7):768-76. doi: 10.1176/appi.ajp.2009.08101604. Epub 2009 May 15. PMID 19448186
- [Background] Taghva A, Oluigbo C, Corrigan J, Rezai AR. Posttraumatic stress disorder: neurocircuitry and implications for potential deep brain stimulation. Stereotact Funct Neurosurg. 2013;91(4):207-19. doi: 10.1159/000343148. Epub 2013 Mar 26. PMID 23548850
- [Background] Taghva A, Silvetz R, Ring A, Kim KY, Murphy KT, Liu CY, Jin Y. Magnetic Resonance Therapy Improves Clinical Phenotype and EEG Alpha Power in Posttraumatic Stress Disorder. Trauma Mon. 2015 Nov;20(4):e27360. doi: 10.5812/traumamon.27360. Epub 2015 Nov 23. PMID 26839865
- [Background] Tanelian, T L; Jaycox, L, eds. (2008). Invisible wounds of war: psychological and cognitive injuries, their consequences, and services to assist recovery. RAND Center for Military Health Policy Research. Santa Monica, CA: RAND Corporation.
- [Background] The Columbia Protocol: About the Protocol. (2016). Retrieved October 24, 2020, from The Columbia Lighthouse Project: Identify Risk, Prevent Suicide: https://cssrs.columbia.edu/the-columbia-scale-c-ssrs/about-the-scale/
- [Background] The Ohio State University Wexner Medical Center. (2020). Ohio State University TBI Identification Method. Retrieved October 23, 2020, from The Ohio State University Wexner Medical Center: https://wexnermedical.osu.edu/neurological-institute/departments-and-centers/research-centers/ohio-valley-center-for-brain-injury-prevention-and-rehabilitation/osu-tbi-id
- [Background] Thomas JL, Wilk JE, Riviere LA, McGurk D, Castro CA, Hoge CW. Prevalence of mental health problems and functional impairment among active component and National Guard soldiers 3 and 12 months following combat in Iraq. Arch Gen Psychiatry. 2010 Jun;67(6):614-23. doi: 10.1001/archgenpsychiatry.2010.54. PMID 20530011
- [Background] Thompson, C., Davies, P., Herrmann, L., Summers, M., & Potter, S. (2016, March). Approaches to establishing validated cut-off scores on the Rivermead Post Concussion Symptoms Questionnaire (RPQ). Brain Injury, 30(5-6), 770.
- [Background] U.S. Department of Veterans Affairs. (2015, December 3). PTSD Checklist for DSM-5 (PCL-5). Retrieved from U.S. Department of Veterans Affairs PTSD: National Center for PTSD: http://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp
- [Background] U.S. Department of Veterans Affairs. (2020, August 10). Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Retrieved 10 19, 2020, from PTSD: National Center for PTSD: https://www.ptsd.va.gov/professional/assessment/adult-int/caps.asp
- [Background] U.S. Department of Veterans Affairs. (2020, June 9). PTSD Checklist for DSM-5 (PCL-5). Retrieved July 13, 2020, from PTSD: National Center for PTSD: https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp
- [Background] United States Army Medical Command. (2014, March 4). OSTG/MEDCOM Policy Memo 14-019. Inpatient and Emergency Department (ED) Aftercare; MEMORANDUM FOR COMMANDERS, MEDCOM REGIONAL MEDICAL COMMANDS. JBSA Fort Sam Houston, Texas, USA.
- [Background] United States Department of Veterans Affairs. (2020, August 10). Combat Exposure Scale (CES). Retrieved October 24, 2020, from National Center for PTSD: https://www.ptsd.va.gov/professional/assessment/te-measures/ces.asp
- [Background] United States Food and Drug Administration. (2012). Guidance for Industry; Suicidal Ideation and Behavior: Prospective Assessment of Occurrence in Clinical Trials (Draft Guidance). Center for Drug Evaluation and Research (CDER). Retrieved October 24, 2020, from https://www.fda.gov/regulatory-information/search-fda-guidance-documents/guidance-industry-suicidal-ideation-and-behavior-prospective-assessment-occurrence-clinical-trials
- [Background] United States Food and Drug Administration. (July 27, 2016). Guidance: Adaptive Designs for Medical Device Clinical Studies. Rockville, MD: U.S. FDA, Center for Devices and Radiological Health, Center for Biologics Evaluation and Research.
- [Background] University of Pittsburgh. (2020, October 23). Measures and Study Instruments. Retrieved from University of Pittsburgh Center for Sleep and Circadian Science: https://www.sleep.pitt.edu/instruments/#psqi
- [Background] Management of Concussion/mTBI Working Group. VA/DoD Clinical Practice Guideline for Management of Concussion/Mild Traumatic Brain Injury. J Rehabil Res Dev. 2009;46(6):CP1-68. No abstract available. PMID 20108447
- [Background] Valenza G, Garcia RG, Citi L, Scilingo EP, Tomaz CA, Barbieri R. Nonlinear digital signal processing in mental health: characterization of major depression using instantaneous entropy measures of heartbeat dynamics. Front Physiol. 2015 Mar 13;6:74. doi: 10.3389/fphys.2015.00074. eCollection 2015. PMID 25821435
- [Background] Van Etten ML, et. al. (1998). Comparative Efficacy of Treatements for Post-traumatic Stress Disorder: A Meta-Analysis. Clin Psychol. Psychother, 5, 126-144.
- [Background] Vasterling JJ, Brailey K, Constans JI, Sutker PB. Attention and memory dysfunction in posttraumatic stress disorder. Neuropsychology. 1998 Jan;12(1):125-33. doi: 10.1037//0894-4105.12.1.125. PMID 9460740
- [Background] Vasterling JJ, Duke LM, Brailey K, Constans JI, Allain AN Jr, Sutker PB. Attention, learning, and memory performances and intellectual resources in Vietnam veterans: PTSD and no disorder comparisons. Neuropsychology. 2002 Jan;16(1):5-14. doi: 10.1037//0894-4105.16.1.5. PMID 11853357
- [Background] Vinck M, Oostenveld R, van Wingerden M, Battaglia F, Pennartz CM. An improved index of phase-synchronization for electrophysiological data in the presence of volume-conduction, noise and sample-size bias. Neuroimage. 2011 Apr 15;55(4):1548-65. doi: 10.1016/j.neuroimage.2011.01.055. Epub 2011 Jan 27. PMID 21276857
- [Background] Wade DT, King NS, Wenden FJ, Crawford S, Caldwell FE. Routine follow up after head injury: a second randomised controlled trial. J Neurol Neurosurg Psychiatry. 1998 Aug;65(2):177-83. doi: 10.1136/jnnp.65.2.177. PMID 9703167
- [Background] Waite, J. C. (2017). Assessing Blinding in Randomized Clinical Trials. Masters Thesis in Mathematics;. California State Polytechnic University. Retrieved from http://dspace.calstate.edu/bitstream/handle/10211.3/196699/WaiteJesse_Thesis2017.pdf?sequence=6
- [Background] Warden D. Military TBI during the Iraq and Afghanistan wars. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):398-402. doi: 10.1097/00001199-200609000-00004. PMID 16983225
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Wassermann EM, Lisanby SH. Therapeutic application of repetitive transcranial magnetic stimulation: a review. Clin Neurophysiol. 2001 Aug;112(8):1367-77. doi: 10.1016/s1388-2457(01)00585-5. PMID 11459676
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Weathers et. al. (2020, March 12). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). [Assessment]. Retrieved March 17, 2020, from U.S. Department of Veterans Affairs: PTSD: National Center for PTSD: www.ptsd.va.gov
- [Background] Weathers, F. W., Blake, D. D., Schnurr, P. P., Kaloupek, D. G., Marx, B. P., & Keane, T. M. (2020, September 29). PTSD: National Center for PTSD. Retrieved 10 19, 2020, from U.S. Department of Veterans Affairs: https://www.ptsd/valgov/professional/assessment/te-measures/life_events_checklist.aspl
- [Background] Wippold FJ 2nd; Expert Panel on Neurologic Imaging. Focal neurologic deficit. AJNR Am J Neuroradiol. 2008 Nov;29(10):1998-2000. No abstract available. PMID 19008324
- [Background] Wobrock T, Guse B, Cordes J, Wolwer W, Winterer G, Gaebel W, Langguth B, Landgrebe M, Eichhammer P, Frank E, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Malchow B, Schneider-Axmann T, Falkai P, Hasan A. Left prefrontal high-frequency repetitive transcranial magnetic stimulation for the treatment of schizophrenia with predominant negative symptoms: a sham-controlled, randomized multicenter trial. Biol Psychiatry. 2015 Jun 1;77(11):979-88. doi: 10.1016/j.biopsych.2014.10.009. Epub 2014 Oct 23. PMID 25582269
- [Background] Wolf EJ, Miller MW, Reardon AF, Ryabchenko KA, Castillo D, Freund R. A latent class analysis of dissociation and posttraumatic stress disorder: evidence for a dissociative subtype. Arch Gen Psychiatry. 2012 Jul;69(7):698-705. doi: 10.1001/archgenpsychiatry.2011.1574. PMID 22752235
- [Background] World Health Organization, editors. (1993). The ICD-10 Classification of Mental and Behavioural Disorders Diagnostic Criteria for Research. Geneva: World Health Organization.
- [Background] Xia G, Gajwani P, Muzina DJ, Kemp DE, Gao K, Ganocy SJ, Calabrese JR. Treatment-emergent mania in unipolar and bipolar depression: focus on repetitive transcranial magnetic stimulation. Int J Neuropsychopharmacol. 2008 Feb;11(1):119-30. doi: 10.1017/S1461145707007699. Epub 2007 Mar 5. PMID 17335643
- [Background] Yehuda R. Post-traumatic stress disorder. N Engl J Med. 2002 Jan 10;346(2):108-14. doi: 10.1056/NEJMra012941. No abstract available. PMID 11784878
- [Background] Yesavage JA, Fairchild JK, Mi Z, Biswas K, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Williams LM, Etkin A, O'Hara R, Georgette G, Beale T, Huang GD, Noda A, George MS; VA Cooperative Studies Program Study Team. Effect of Repetitive Transcranial Magnetic Stimulation on Treatment-Resistant Major Depression in US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Sep 1;75(9):884-893. doi: 10.1001/jamapsychiatry.2018.1483. PMID 29955803
- [Background] Ziemann U. TMS and drugs. Clin Neurophysiol. 2004 Aug;115(8):1717-29. doi: 10.1016/j.clinph.2004.03.006. PMID 15261850
- [Background] Ziemann U, Reis J, Schwenkreis P, Rosanova M, Strafella A, Badawy R, Muller-Dahlhaus F. TMS and drugs revisited 2014. Clin Neurophysiol. 2015 Oct;126(10):1847-68. doi: 10.1016/j.clinph.2014.08.028. Epub 2014 Dec 4. PMID 25534482
- [Background] Zwanzger P, Ella R, Keck ME, Rupprecht R, Padberg F. Occurrence of delusions during repetitive transcranial magnetic stimulation (rTMS) in major depression. Biol Psychiatry. 2002 Apr 1;51(7):602-3. doi: 10.1016/s0006-3223(01)01369-5. PMID 11950462